CLINICAL TRIAL: NCT00484042
Title: Activation of Polyamine Catabolism in Patients With Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Other Study IDs: R06025
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatitis; Polyamines
Keywords: pancreatitis; polyamine; cytokine
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Polyamines are essential compounds in all mammalian tissues. If tissue spermidine/spermine levels, however, dramatically decrease, the cellular survival is severely endangered. Transgenic animals, where the homeostasis of cellular polyamines can be disturbed and tissue spermidine/spermine levels are decreased, acute pancreatitis evolves, indicating pancreas to be one of the most vulnerable organs for tissue polyamine catabolism. On the other hand, our own data suggests that also in other models of acute experimental pancreatitis pancreatic polyamines are changed depending on the severity of pancreatitis in such a way that the more severe pancreatitis the lower are the pancreatic polyamine levels. Minor changes were observed also in rats undergoing sham operation only. In addition of pancreatic enzymes, inflammatory mediators are also involved in the pathophysiology of the disease. CRP, IL-6, IL-8, IL-10 and Procalcitonin are useful in predicting the severity of the disease, combination of IL-6 and IL-10 at admission can predict organ failure with sensitivity of 95 %, specificity of 88 %.

Hypothesis: Similar to experimental pancreatitis, blood polyamine changes are associated with acute pancreatitis also in the man. These changes are dependent on the severity of pancreatitis, but not on the etiology of pancreatitis. The changes are specific to acute pancreatitis compared with other intra-abdominal emergencies. The changes observed return to baseline during recovery. Furthermore, we assume that blood polyamine negatively correlates with IL-6, IL-8, and procalcitonin, and positively with IL-10.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as acute pancreatitis.
* Patients who are diagnosed as either of gallstone, duodenal ulcer or bleeding, gastric ulcer or bleeding, irritable bowel syndrome, hernia, diverticulitis, retrocecal appendicitis with non-pancreatic acute abdominal pain.

Exclusion Criteria:

* Patients who underwent operation
* Patients who underwent recurrent acute pancreatitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-01; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isto H Nordback, M.D., Principal Investigator — Tampere University Hospital